CLINICAL TRIAL: NCT02472002
Title: Mesenchymal Stem Cell Administration in the Treatment of Coronary Graft Disease in Heart Transplant Patients
Acronym: MESHT
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Contamination of the Pitié-Salpêtrière biotherapy laboratory
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P 100102
Record Dates: First submitted 2015-06-01; First posted 2015-06-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Coronary Disease; Heart Transplant
Keywords: Transplant coronary diseases; Mesenchymal cell therapy; Administration of CSM by NOGA system; Coronary disease in heart transplant patients
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesenchymal cell therapy (Experimental)
  Interventions: Biological: Mesenchymal cell therapy

INTERVENTIONS:
Biological: Mesenchymal cell therapy — Name of the experimental cell preparation: Concentrated mesenchymal stem cells (MSCs) derived from autologous bone marrow
  * Registry Type: autologous
  * Qualitative and quantitative composition of the finished product: The product is a cell suspension consisting of mesenchymal stem cells (MSC) 40 x 106 MSC / ml suspended in human albumin (ALBUNORM ® 5% OCTAPHARMA France).
  * Route of administration: endomyocardial injection
  * Dose administered: 120-140 x106 MSC (mesenchymal stem cells)

SUMMARY:
MES-HT is a pilot multicenter prospective study conducted in transplant patients who developed severe coronary vasculopathy. A preparation of autologous mesenchymal cells of bone marrow is administered by endomyocardial injection, guided by the Noga® cardiac mapping system.

The main objective is to determine the effect of the administration of autologous mesenchymal cells of the bone marrow by intramyocardial injection on myocardial perfusion in cardiac transplant patients with severe coronary vasculopathy.

DETAILED DESCRIPTION:
MES-HT is a phase 1-2 multicenter pilot prospective study conducted on 14 heart transplant patients who developed severe coronary vasculopathy, in the aim to assess the effect on myocardial perfusion of the intramyocardial administration by percutaneous way of autologous mesenchymal stem cells derived from the bone marrow.

The main objective is to show improvement in myocardial perfusion in a non-randomized and uncontrolled pilot study, before considering a randomized controlled study. The administration of intra myocardial cells using the NOGA system was carried out to date with more than 1,000 patients and is considered feasible and safe. However, the investigators will assess very carefully the feasibility and safety of this invasive approach.

The primary endpoint is the improvement of myocardial perfusion measured by MRI after endomyocardial injection of mesenchymal cells by percutaneous way, guided by the NOGA system.

The secondary endpoints are the feasibility and safety of this administration, changes in ejection fraction measured by contrast echocardiography, changes in other MRI cardiac parameters (left ventricular volumes , intramyocardial fibrosis), the oxygen consumption during exercise, myocardial perfusion measured by SPECT. Other secondary endpoints are the evolution of the immune status, and histological criteria of myocardial biopsy.

Once the mapping performed, preparation is injected through another catheter (MYOSTAR injection catheter) which will also be guided by the Noga® system. This catheter may be positioned on the regions of interest (viable ischemic areas) and allow the injection of the quantity of CSM (40 million / ml) in 10 to 12 different injection points and injection volumes 0.3 ml for a total dose of 120 to 144 million cells.

After each injection procedure, patients are monitored for 48 hours minimum clinically and under continuous ECG monitoring to detect possible arrhythmias. A troponin dosage is done after 6 H, and after 24 and 48 hours. An echocardiogram is performed immediately after the procedure and before the release to 48 H.

A clinical evaluation will be made after the patient is discharged at 1 month (clinical examination + Holter + echocardiography), 3 months (examination), 6 months (clinical examination, Holter, echocardiography, cardiac MRI, test of effort with measurement of VO2, effort myocardial tomoscintigraphy and for patients from Pitie-Salpetriere hospital, Rubidium 82 by positron emission tomography) and 12 months (examination). Myocardial biopsy and a control coronary angiography will be only performed within 12 months in accordance with the practice of the teams.

Patients will benefit from a biological monitoring which provides for the monitoring of immune response. This immuno-monitoring is to assess the possible influence of the injection of mesenchymal cells on immunological tolerance mechanisms. It will be implemented in the balance sheets of cardiac tissue at the waning annual biopsies and peripheral blood samples on inclusion, 48 hours after injection and at 1 month, 3 months and 6 months.

The limiting toxicity is defined as the occurrence at one month of a serious adverse effect related to the protocol , requiring an hospitalization or being able to be life-threatening , or like abundant pericardial effusion requiring pericardial drainage, bleeding complications requiring blood cell transfusion or surgery, stroke constituted, sepsis or septic shock, cardiogenic shock, severe ventricular rhythm refractory death.

All patients are followed for one year.

ELIGIBILITY:
Inclusion criteria :

1. Cardiac transplant patient whatever is his initial pathology
2. Coronary vasculopathy grade 3 (CAV3) defined by:

   Stenosis > 50% of common-core (CT) or stenosis >70% of at least 2 or 3 main coronary arteries or stenosis > 70% on secondary branches of 3 territories.

   Coronary vasculopathy grade 1 or 2 (CAV 1 or 2) associated with FELV (FEVG) dysfunction <45% or abnormality of completion of restrictive type.
3. Defect of drip on at least 2 segments/17 in stress MRI.
4. Fraction of ejection LV<50 measured on ultrasound examination or confusion of diastolic function defined by a restrictive mitral steam (E/A > 2 or E/A between 1 and 2 and deceleration time E < 150 ms) or left ventricular diastolic pressure measured during coronarography >16mg Hg .
5. Without sign of acute rejection at the time of inclusion.
6. Under an optimal medical treatment
7. Patient who have given his enlightened and signed consent

Exclusion criteria :

1. Patients <18 ou >80 years
2. Acute coronary syndrome or revascularisation in the 3 last months
3. Acute cardiac rejection in the 3 last months
4. Atrial fibrillation
5. Claustrophobia or contraindication to MRI (ex:pace-maker), to contrast injection or adenosine.
6. Presence of a thrombus in the left cavities detected by ultra-sound examination or MRI realized before the injection..
7. Pregnant or breast-feeding woman
8. Woman old enough to reproduction without effective means of contraception during its participation in the study
9. Patient benefiting from a legal protective measure
10. HIV positive
11. Not membership in a national save insurance (beneficiary or legal successor)
12. Patients undergoing others biomedical research
13. Patient not understanding the procedure bound to the protocol
14. Bad adhesion to the protocol suspected by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
myocardial perfusion measured in MRI. | 6 months

SECONDARY OUTCOMES:
complications of catheterization | 6 months
complications of endomyocardial injection | 6 months
systolic function | 6 months
diastolic function | 6 months
immunomodulation induced MSCs in the blood | 6 months
immunomodulation induced MSCs in myocardial biopsy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Isnard, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Département de cardiologie du Pr Michel KOMADJA, Paris, France